CLINICAL TRIAL: NCT04082299
Title: Immune Response Following Tdap Vaccination in Pregnant vs. Non Pregnant Women
Brief Title: Immune Response followingTdap Vaccine in Pregnancy
Status: Completed | Type: Observational
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0079-19-HYMC
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Diphtheria-Tetanus-acellular Pertussis Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood for Immunoglobulin G analysis, umbilical blood and mother milk.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pregnant women: pregnant women expected to be vaccinate with Tdap vaccine during their 3th trimester
- Non pregnant women: Non pregnant women expected to be vaccinate with Tdap vaccine

SUMMARY:
Pregnancy involves changes in immune response. The investigators aim to evaluate the immune response to Tdap in pregnancy in comparison to non pregnant women usig proteomics and gene sequencing.

DETAILED DESCRIPTION:
Many vaccine-preventable diseases, like influenza, pertussis, and tetanus cause substantial morbidity and mortality in pregnant women, newborns and infants. Immunization during pregnancy has the potential to provide protection to the newborn and infant by the transplacental transfer of vaccine-specific maternal antibodies. However, the immunobiology underlying immunization during pregnancy, that leads to the protection of the newborn are not understood. Current vaccine formulations were designed for and tested in non-pregnant populations; yet substantial immune modulations take place during different stages of pregnancy and potentially can impact the humoral response following maternal immunization. The investigators thus have insufficient data on quantity and quality of the immune response during pregnancy and how this relates to immunity provided from the mother to the newborn. First, The investigators hypothesize that the nature and breadth of the humoral immune response following vaccination differs in pregnant and non-pregnant vaccinees. Next, The investigators hypothesize that the vaccine-specific antibodies that cross the placenta, comprise distinct repertoire features thus, the placenta functions as a differential barrier for antibody transfer. To test these hypotheses, The investigators will use proteomic and genomic/transcriptomic measurements of antibody repertoires in the maternal and cord blood compartments. The measurements will be based on antibody clonal diversity/frequency, V(D)J germline usage and SHM, where we expect to find changes in i) vaccine-specific B cell frequency, antibody clonal diversity, germline usage and SHM in pregnant women and ii) distinct repertoire features in the transplacental vaccine-specific antibody compartment compared the maternal compartment. The investigators will utilize deep sequencing and proteomic technologies to provide, for the first time, insight into the immunobiology of a promising intervention aimed to prevent early life infectious morbidity and mortality and establish new research avenues for vaccine research in vulnerable populations.

ELIGIBILITY:
Inclusion Criteria for pregnant women (cohort 1):

* age between 18-45 years
* pregnant women who expected to have Tdap vaccine
* Informed Consent Form signature

Inclusion Criteria for non pregnant women (cohort 2):

* age between 18-45 years
* non pregnant women who expected to have Tdap vaccine
* Informed Consent Form signature

Exclusion Criteria (cohort 1 and 2):

* any background immune diseases- autoimmune conditions or cancer.
* women who take immunosuppressive/ immunomodulatory medications
* a patient has received Tdap vaccine in 6 months prior to study entry.
* no will to signed the Informed Consent Form.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant and non pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

PRIMARY OUTCOMES:
Immune response following Tdap vaccine | 4 months
  Characterization of immune response following Tdap vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Rinat Gabbay-Benziv, Dr, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe medical center, Hadera, Israel